CLINICAL TRIAL: NCT07134205
Title: A Randomized, Open-label, Multicenter Phase III Clinical Study of JMT101 in Combination With Irinotecan in Third-line and Beyond Treatment of Metastatic Colorectal Cancer
Brief Title: The Study of JMT101 Combined With Irinotecan as a ≥3rd-Line Treatment in Metastatic Colorectal Cancer
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMT101-017
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Colorectal Cancer (mCRC)
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Irinotecan; regorafenib

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- JMT101 + Irinotecan (Experimental): JMT101, 6 mg/kg, Irinotecan, 180mg/m^2, administered by IV infusion once every two weeks (one treatment cycle is 4 weeks).
  Interventions: Drug: JMT101; Drug: Irinotecan
- Standard of care (Active Comparator): 28 day for one cycle.
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: JMT101 — JMT101, 6 mg/kg, administered by IV infusion once every two weeks (one treatment cycle is 4 weeks).
  Arms: JMT101 + Irinotecan
Drug: Irinotecan — Irinotecan, 180mg/m^2, administered by IV infusion once every two weeks (one treatment cycle is 4 weeks).
  Arms: JMT101 + Irinotecan
Drug: Regorafenib — Regorafenib, 160 mg, taken orally once daily for the first 21 days of each 28-day cycle.
  Arms: Standard of care

SUMMARY:
This is a randomized, open-label, multicenter, phase III clinical study. The aim is to evaluate the efficacy of JMT101 in combination with irinotecan in the third-line and beyond treatment of Metastatic Colorectal Cancer.

DETAILED DESCRIPTION:
This trial is conducted in patients with refractory metastatic colorectal cancer that has progressed after second-line or higher standard therapy. Eligible patients are randomized into two arms in a 1:1 ratio to receive JMT101 in combination with irinotecan or standard of care until disease progression, unacceptable toxicity or withdrawal of consent by the patient.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ranged from 18 to 75 years old (inclusive), regardless of gender;
* 2. Pathological diagnosis as metastatic colorectal adenocarcinoma, with RAS and BRAF wild-type and non-dMMR/MSI-H;
* 3. Tumor tissue available for central laboratory testing;
* 4. Metastatic colorectal cancer with disease progression after 2nd line treatment; previously received standard chemotherapy based on fluorouracil, oxaliplatin, irinotecan; patients are allowed to previously receive EGFR and/or VEGF inhibitors, but not allowed to previously receive regorafenib, fruquintinib;
* 5. Measurable disease according to RECIST1.1;
* 6. Eastern Cooperative Oncology Group (ECOG) score 0-1 points;
* 7. Life expectancy ≥3 months
* 8. Adequate main organs and bone marrow function.
* 9. Patients must give informed consent to this study before the experiment and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1. Participants who have been systematically treated with an EGFR inhibitor (such as cetuximab) within 4 months prior to the first dose of study drug.
* 2. Central nervous system metastasis or meningeal metastasis;
* 3. Patients with high risk of bleeding due to tumor invasion of important arteries;
* 4. Uncontrolled or requiring repeated drainage of pleural effusion, pericardial effusion, or abdominal effusion;
* 5. The adverse reactions of previous anti-tumor treatments (including radiotherapy) have not yet recovered to CTCAE 5.0 evaluation ≤ level 1;
* 6. Diagnosed as a second primary malignant tumor within 5 years prior to the first administration of the study drug;
* 7. Have received anti-tumor treatments such as chemotherapy, biological therapy, targeted therapy, etc. within 21 days before the first dose of the study drug; radiotherapy within 2 weeks before the first dose of the study drug; Chinese medicine or Chinese patent medicine with anti-tumor effect within 1 week before the first dose of the study drug;
* 8. Have received a live viral vaccine or live-attenuated vaccine within 28 days before the first dose of study drug or plan to receive it during the study;
* 9. Use of immunosuppressive medications within 14 days prior to the first dose of study drug;
* 10. Those who use strong CYP3A4 inducers within 14 days before the first administration of the study drug, or those who use strong CYP3A4 inhibitors or strong UGT1A9 inhibitors within 2 week, or those who cannot suspend the use of the above drugs during the study;
* 11. Have received radiation therapy or other localized palliative treatment within 14 days before the first dose of study drug;
* 12. Have undergone major surgery (excluding needle biopsy) or suffered severe traumatic injury within 28 days before the first dose of study drug;
* 13. Have a history of serious cardiovascular disease;
* 14. Previous or current presence of interstitial pneumonia/lung disease;
* 15. History of autoimmune diseases;
* 16. A history of immunodeficiency, including HIV testing positive, or having other acquired or congenital immunodeficiency diseases, or having a history of organ transplantation;
* 17. Have infectious diseases requiring systemic anti-infective treatment;
* 18. Active hepatitis B; hepatitis C infection; syphilis infection, active tuberculosis;
* 19. Known presence of hypersensitivity or intolerance to any component of EGFR monoclonal antibody, irinotecan hydrochloride injection, regorafenib and its excipients;
* 20. Women during lactation or pregnancy; women with fertility tested positive for blood pregnancy within 7 days prior to enrollment in the trial;
* 21. Any male and female patients with fertility who refuse to use effective contraceptive methods throughout the entire trial period and within six months after the last administration;
* 22. Other conditions that, in the opinion of the investigator, may affect the safety or compliance of drug treatment in this study, including but not limited to: psychiatric disorders, any severe or uncontrollable diseases, etc.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 3 years
  defined as the time from randomization to the first occurrence of disease progression as determined by the BIRC with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 2 years
  determined by the BIRC and investigator with use of RECIST v1.1
Disease Control Rate (DCR) | Up to approximately 2 years
  determined by the BIRC and investigator with use of RECIST v1.1
Duration of response (DOR) | Up to approximately 2 years
  determined by the BIRC and investigator with use of RECIST v1.1
Progression-free Survival (PFS) | Up to approximately 2 years
  defined as the time from randomization to the first occurrence of disease progression as determined by the investigator with use of RECIST v1.1 or death from any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 5 years
  Duration from the date of initial treatment to the date of death due to any cause.
Incidence and severity of AEs | Up to approximately 2 years
  Incidence and severity of adverse events (AE). Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
Serum concentration of JMT101 | Up to approximately 2 years
  Serum concentration and immunogenicity of JMT101
Serum immunogenicity of JMT101 | Up to approximately 2 years
  Immunogenicity of JMT101
To be assessed by European Quality of Life Five Dimensions Questionnaire (EQ-5D-5L). | Up to approximately 2 years
  use EORTC QLQ-C30 questionnaire and the EQ-5D-5L questionnaire
Drug resistance | Up to approximately 2 years
  Gene Variations Detected by ctDNA and Drug Resistance Biomarkers